CLINICAL TRIAL: NCT06967883
Title: The Relationship Between Ultrasonographic Measurements of Cervical Multifidus and Longus Colli Muscles and Balance in Male Patients With Ankylosing Spondylitis:Controlled Study
Brief Title: Ultrasound Assessment of Neck Muscles and Balance in Male Patients With Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ISTPMRTRH2024-80
Record Dates: First submitted 2025-02-23; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Ankylosing Spondylitis; Balance Assessment; Balance; Spondylarthropathies; Spondylitis, Ankylosing
Keywords: ankylosing spondylitis; balance; deep cervical muscles
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthropathies; Spondylitis | interventions — Postural Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis Group: Male patients aged 18-65 years diagnosed with Ankylosing Spondylitis according to the Modified New York Criteria, under regular follow-up at Istanbul Physical Medicine and Rehabilitation Rheumatology Clinic.
  Interventions: Diagnostic Test: Ultrasonographic assessment of Cervical Multifidus and Longus Colli Muscle Thickness, Postural Balance and Limit of Stability using the balance platform,Cervical Flexion and Extension Strength
- Control Group: Age-matched healthy male volunteers aged 18-65 years with cognitive ability sufficient to understand test instructions.
  Interventions: Diagnostic Test: Ultrasonographic assessment of Cervical Multifidus and Longus Colli Muscle Thickness, Postural Balance and Limit of Stability using the balance platform,Cervical Flexion and Extension Strength

INTERVENTIONS:
Diagnostic Test: Ultrasonographic assessment of Cervical Multifidus and Longus Colli Muscle Thickness, Postural Balance and Limit of Stability using the balance platform,Cervical Flexion and Extension Strength — Intervention Description
  Participants in both groups will undergo ultrasonographic measurement of cervical multifidus and longus colli muscle thickness. Postural sway, Limits of Stability (LOS), and a 6-direction balance test (ABC-6) will be assessed using the HUR SmartBalance BTG4 platform under stable and unstable conditions with eyes open and closed. Functional balance will be evaluated with the Berg Balance Scale (BBS), Timed Up and Go (TUG) Test, and Single-Leg Stance Test. Isometric cervical flexion and extension strength will be measured bilaterally using a hand-held dynamometer. Ankylosing Spondylitis patients will additionally complete BASFI, BASMI, BASDAI, and ASQoL questionnaires.

SUMMARY:
The aim of this study is to evaluate the relationship between ultrasonographic measurements of the cervical muscles and balance parameters in patients diagnosed with ankylosing spondylitis (AS)

DETAILED DESCRIPTION:
This study aims to investigate the relationship between cervical multifdus and longus Colli muscles and balance function in male patients diagnosed with Ankylosing Spondylitis (AS) according to the Modified New York Criteria. A total of 38 AS patients under regular follow-up at the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital Rheumatology Clinic, along with 38 age-matched healthy male volunteers, will be included.

Ultrasonographic Imaging will be performed to assess the thickness and of the cervical multifidus and longus colli muscles.The HUR SmartBalance BTG4 (HUR-Labs Oy, Kokkola, Finland) balance platform will be used to measure postural sway, weight distribution, and the limit of stability (LOS) through a computerized system.The Berg Balance Scale (BBS), The Timed Up and Go (TUG) test,The Single-Leg Stance Test will be conducted, measuring the ability to maintain posture while standing on one leg. Disease Activity and Functional Assessment in AS Patients will be conducted by using The Bath Ankylosing Spondylitis Functional Index (BASFI), The Bath Ankylosing Spondylitis Metrology Index (BASMI) Additionally, the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be used to measure disease activity and quality of life will be assessed with Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL).Cervical Muscle Strength Measurement will be performed using a hand-held dynamometer, which will objectively assess isometric cervical flexion and extension strength.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosed with Ankylosing Spondylitis according to the Modified New York Criteria (for patient group).
* Cognitive ability sufficient to understand and follow test instructions.

Exclusion Criteria:

* Orthopedic disorders affecting the spine or lower limbs.
* Cardiovascular disorders.
* Neurological disorders.
* Visual or auditory impairments.
* History of surgery involving the spine or lower limbs.
* Psychiatric disorders.
* Cognitive impairment.
* Clinical signs or symptoms of cervical radiculopathy.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Istanbul Physical Medicine and Rehabilitation Rheumatology Clinic, where they are under regular follow-up for Ankylosing Spondylitis (AS). The healthy control group will consist of hospital employees who meet the inclusion criteria and have no history of AS or other musculoskeletal disorders
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Mean Bilateral Thickness of Cervical Multifidus Muscle Assessed by Ultrasonography | baseline
  Bilateral measurement of cervical multifidus muscle thickness using musculoskeletal ultrasound imaging. Results will be reported in millimeters (mm). Data will be summarized as mean ± standard deviation.
Mean Bilateral Thickness of Cervical Longus Colli Muscle Assessed by Ultrasonography | baseline
  Bilateral measurement of cervical longus colli muscle thickness using musculoskeletal ultrasound imaging. Results will be reported in millimeters (mm). Data will be summarized as mean ± standard deviation.
Limits of Stability (LOS) Test | baseline
  The Limits of Stability (LOS) test will be conducted using the HUR SmartBalance platform. Participants will be asked to lean maximally forward, backward, to the right, and to the left, each for a duration of 8 s without lifting the sole and heel of the foot or correcting their feet. Using these methods, the individual's stability limits will be tested in four directions. The LOS score quantifies the subject's ability to voluntarily control posture within their stability limits. The leaning angle is based on the person's height and how far the center of pressure move from the normal position. A lower LOS score indicates impaired postural control and balance performance.

SECONDARY OUTCOMES:
Sway Area on Balance Platform | baseline
  Postural sway area measured as 90% confidence ellipse (C90) using the HUR SmartBalance BTG4 platform. Results will be reported in square millimeters (mm²). Data will be summarized as mean ± standard deviation.
Romberg Quotient | baseline
  Ratio of sway areas between eyes-open and eyes-closed conditions. Results will be reported as a dimensionless ratio. Data will be summarized as mean ± standard deviation.
Trace Length on Balance Platform | baseline
  Total trace length of center of pressure movement during static standing, measured using the HUR SmartBalance BTG4 platform. Results will be reported in millimeters (mm). Data will be summarized as mean ± standard deviation.
Medio-Lateral (ML) Sway Range | baseline
  Range of center of pressure displacement in the medio-lateral direction during standing balance tests. Results will be reported in millimeters (mm). Data will be summarized as mean ± standard deviation.
Anterior-Posterior (AP) Sway Range | baseline
  Range of center of pressure displacement in the anterior-posterior direction during standing balance tests. Results will be reported in millimeters (mm). Data will be summarized as mean ± standard deviation.
Average Sway Velocity | baseline
  Average sway velocity calculated by dividing the total trace length by the duration of the test. Results will be reported in millimeters per second (mm/s). Data will be summarized as mean ± standard deviation.
Timed Up and Go (TUG) Test Duration | baseline
  ime required to complete the Timed Up and Go (TUG) test. Results will be reported in seconds (s). Data will be summarized as mean ± standard deviation.
Berg Balance Scale Total Score | baseline
  Total score on the Berg Balance Scale (range 0-56 points) assessing functional balance. Results will be reported as a unitless total score. Data will be summarized as mean ± standard deviation.

OTHER OUTCOMES:
Isometric Cervical Flexion and Extension Strength Measured by Hand-Held Dynamometer | baseline
  Isometric strength of cervical flexor and extensor muscles assessed bilaterally using a hand-held dynamometer. Results will be reported in Newtons (N). Data will be summarized as mean ± standard deviation.
Short Version of the Activities-Specific Balance Confidence Scale (ABC-6) Score | baseline
  Balance confidence will be assessed using the Short Version of the Activities-Specific Balance Confidence Scale (ABC-6), where participants rate their confidence in performing six common daily activities without losing balance. Each item is scored from 0 (no confidence) to 100 (complete confidence). The final score will be reported as the mean of all item scores. Results will be summarized as mean ± standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Paker, MD, Prof., Study Director — Istanbul Physical Medicine and Rehabilitation Training Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Trainig and Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozen T, Tonga E, Polat MG, Bayraktar D, Akar S. Cervical proprioception accuracy is impaired in patients with axial spondyloarthritis. Musculoskelet Sci Pract. 2021 Feb;51:102304. doi: 10.1016/j.msksp.2020.102304. Epub 2020 Nov 16. PMID 33227676
- [Background] Turk E, Yurdakul FG, Guler T, Bodur H. Posture, balance and gait in axial spondyloarthritis: a case-control study. Rheumatol Int. 2024 Nov;44(11):2527-2538. doi: 10.1007/s00296-024-05710-5. Epub 2024 Sep 4. PMID 39230687
- See also: Sonographic Comparison of Neck Extensor Muscle Thickness of Ankylosing Spondylitis and Non-radiographic Axial Spondyloarthritis Patients with Healthy Volunteers — https://www.thieme-connect.com/products/ejournals/pdf/10.1055/a-1853-9489.pdf